CLINICAL TRIAL: NCT06087861
Title: Phase 2 5-Day Preoperative Radiation for Soft Tissue Sarcoma
Brief Title: 5-Day Preoperative Radiation for Soft Tissue Sarcoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-71865; NCI-2024-00868 (Registry Identifier: NCI- Clinical Trials Reporting Program)
Record Dates: First submitted 2023-10-11; First posted 2023-10-18 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- External beam radiotherapy (Experimental): Patients will receive treatment with external beam radiotherapy at a total of 30 Gy delivered over five fractions delivered daily.
  Interventions: Radiation: External Beam Radiotherapy

INTERVENTIONS:
Radiation: External Beam Radiotherapy — Radiation will be delivered by external beam techniques to the tumor and areas of possible microscopic disease at a dose of 30 Gy divided into 5 equal fractions of 6 Gy (administered over a total of 5 to 10 business day

SUMMARY:
The purpose of this study is to examine the safety and efficacy of an abbreviated course of preoperative radiation, given over five days, for patients with soft tissue sarcoma of the extremity, trunk or retroperitoneum. This is in contrast to standard preoperative radiation, which is given over 25 days.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed soft tissue sarcoma of the extremity, trunk or retroperitoneum.
2. Has been offered preoperative radiation and surgery as part of standard-of-care treatment
3. Age ≥ 18
4. KPS ≥ 70 or ECOG 0 to 2
5. Life expectancy ≥ 6 months
6. If a woman is of childbearing potential, a negative serum or urine pregnancy test must be documented.
7. Ability to understand and the willingness to personally sign the written IRB approved informed consent document.

Exclusion Criteria:

1. History of prior radiation to the area to be treated.
2. Active use of other anti-cancer investigational agents.
3. Planned use of concurrent chemotherapy, targeted therapy, or immunotherapy with radiation therapy (defined as the time interval starting 1 week before the first and last fraction of radiation therapy and surgery).
4. Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-10-06 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Post-operative Complication Rate | 120 days after surgery
  Rate of post-operative complications.

SECONDARY OUTCOMES:
Local Recurrence Rate | 2 years and 5 years after surgical resection
  Rate of local recurrence, including in-field, borderline and out-field recurrences

CONTACTS AND LOCATIONS:
Overall Officials: Anusha Kalbasi, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States